CLINICAL TRIAL: NCT04814602
Title: Single-dose Pharmacokinetic (PK) Assessment of Oral Proglumide in Those With Hepatic Impairment
Brief Title: Single-dose PK Assessment of Oral Proglumide in Those With Hepatic Impairment
Acronym: HIPK
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3464
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-07

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Proglumide

STUDY DESIGN:
Intervention Model Description: open labeled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Healthy controls Proglumide 400 mg given once by mouth
  Interventions: Drug: Proglumide
- Hepatic Impaired (Experimental): Cirrhosis Child-Pugh A and B Proglumide 400 mg given once by mouth
  Interventions: Drug: Proglumide

INTERVENTIONS:
Drug: Proglumide — CCK receptor antagonist
  Other Names: Milid

SUMMARY:
Proglumide is an oral cholecystokinin (CCK) receptor antagonist that has been shown in non-clinical studies to reverse hepatic fibrosis and decrease the incidence of hepatocellular carcinoma (HCC). Because of these potential beneficial properties, proglumide may be useful in decreasing the fibrosis and risk for HCC in those with cirrhosis. Although proglumide is safe in those with normal hepatic function, the pharmacokinetics have not been established in those that are hepatic impaired. The purpose of this study is to analyze proglumide blood levels and excretion in subjects with cirrhosis compared to health controls.

DETAILED DESCRIPTION:
The purpose of this study is to measure blood levels of proglumide after a single oral dose (400 mg) over a period of time and compare the blood levels to those with normal hepatic function (N=4) to determine if there is delayed metabolism and clearance of proglumide in those with hepatic impairment (HI) (N=8). Eligible subjects will provide a baseline blood and urine sample prior to ingesting proglumide 400 mg po. Blood will be collected from an intravenous catheter after ingestion at the following intervals: 1 hr, 3 hrs, 5 hrs, 7 hrs and 24 hr (± 4-5 hours). After 3 hrs and 5 hrs subjects will provide a urine sample. Samples will be analyzed by Mass Spectometry. Proglumide blood and urine levels in ng/ml will be plotted over time and the Cmax (peak plasma concentration), Tmax (time to reach Cmax) and T1/2 (elimination half time) calculated for each subject and compared to that of 4 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis previously confirmed by one of the following: Liver biopsy, FibroScan, FibroSure, MR-Elastography, or nodular liver on radiographic imaging like CT or MRI. Child-Pugh classification A (N=4) and Child-Pugh classification B (N=4)

Exclusion Criteria:

* Those that are Child-Pugh classification C cirrhosis
* gastrointestinal bleeding from esophageal varices within 6 months
* Chronic kidney disease with Estimated glomerular filtration rate (eGFR of < 90 mL/min/1.73m2)
* hepatic encephalopathy
* those that have had an organ transplant
* active hepatitis C, active hepatitis B, and those with HIV disease

  * Adults unable to consent
  * Individuals who are not yet adults (infants, children, teenagers)
  * Pregnant women
  * Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Proglumide blood levels in hepatic impaired subjects | 24 hours
  Proglumide levels in ng/ml in cirrhosis subjects compared to healthy controls

SECONDARY OUTCOMES:
Urinary excretion of proglumide | 24 hours
  Measurement of proglumide in urine after single does ingestion in cirrhosis compared to healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Jill P Smith, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be published and placed on clinicaltrials website